CLINICAL TRIAL: NCT06512584
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of PJ009 in Patients with Short Bowel Syndrome Requiring Parenteral Nutrition
Brief Title: Efficacy and Safety of PJ009 in Patients with Short Bowel Syndrome Requiring Parenteral Nutrition
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chongqing Peg-Bio Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQPJ-PJ009-III
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Glucagon-Like Peptide 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PJ009 (Experimental): subcutaneous injections, 0.05 mg/kg once daily
  Interventions: Drug: PJ009
- PJ009 Placebo (Placebo Comparator): subcutaneous injections, once daily
  Interventions: Drug: PJ009 Placebo

INTERVENTIONS:
Drug: PJ009 — subcutaneous injections, 0.05 mg/kg once daily
  Other Names: Glucagon-Like Peptide 2 (GLP-2) analogue
  Arms: PJ009
Drug: PJ009 Placebo — subcutaneous injections, once daily
  Other Names: GLP-2 analogue Placebo
  Arms: PJ009 Placebo

SUMMARY:
The main aim of this clinical trial is to assess the efficacy and safety of PJ009 in patients aged ≥14 with short bowel syndrome (SBS) requiring parenteral nutrition. The main questions it aims to answer are:

* How effective is PJ009 in treating short bowel syndrome?
* Is PJ009 safe in these patients? Researchers will compare PJ009 to a placebo (a look-alike substance that contains no drug) to see if PJ009 works to treat SBS.

Participants will

* Receive daily subcutaneous injections of PJ009 or placebo according to weight for 24 weeks, and then the participants receive placebo will be switched to receive PJ009 for another 12 weeks, while participants receive PJ009 continued the same treatment until the end of 36 weeks,
* Visit the clinic at the end of week 1(w1), w2, w4, w8, w12, w16, w20, w24, w30 and w36 for assessment,
* Keep a diary of the amount of their parenteral nutrition/ intravenous fluids (PN/IV), enteral nutrition and urine volume.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled clinical study, aiming to evaluate the efficacy, safety, immunogenicity and pharmacokinetic of PJ009 in patients with short bowel syndrome requiring parenteral nutrition, using placebo as a control.

The trial is divided into 3 periods. Period 1 of this trial is the screening, optimization (if applicable, up to 8 weeks) and stabilization (4-8 weeks) period. At the end of the stabilization period, a baseline enrollment evaluation will be performed, and all eligible participants will enter the 24 weeks of double-blind treatment period (period 2). Period 3 is a 12-week open label extension to period 2. Safety follow-up assessments will be performed 4 weeks after the last dose in treatment period 3.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged ≥ 14 years;
2. SBS patients dependent on PN/IV support for at least 6 consecutive months due to major intestinal resection;
3. At least 3 PN/IV support sessions per week are required 1 week before screening or 2 weeks before baseline;
4. Be on stable PN/IV support for at least 4 consecutive weeks before administration;
5. For subjects with a history of Crohn's disease (CD), clinical assessment of remission for at least 12 weeks prior to administration;
6. Be able to understand and provide signed informed consent, for those under 18 years old, the guardian should also sign the informed consent;
7. Be able to complete experiments in accordance with the protocol.

Exclusion Criteria:

1. Have used teduglutide in the past or may be allergic to teduglutide or its components;
2. Have used natural GLP-2 or its analogs, human growth hormone or its analogs within 6 months before screening;
3. Have used glutamine, octreotide, GLP-1 analogs or dipeptidyl peptidase-IV inhibitors within 30 days before screening;
4. With active Crohn's disease or those who need to change biological therapy within 6 months before screening;
5. With active inflammatory bowel disease (IBD) or IBD patients who have received immunosuppressant therapy changes in the past 3 months;
6. With unstable absorption due to cystic fibrosis, untreated megacolon disease or known DNA abnormalities (such as familial adenomatous polyposis, Fanconi syndrome);
7. With clinically obvious intestinal obstruction or active stenosis within 6 months before screening;
8. Have undergone major gastrointestinal surgical intervention within 3 months before screening, such as continuous transverse enteroplasty or other intestinal lengthening surgery (esophageal intubation or endoscopic surgery is allowed);
9. Severe active, uncontrolled, untreated systemic diseases (such as cardiovascular, respiratory, renal, infectious, endocrine, liver or central nervous system diseases, etc.);
10. Have malignant tumors within 5 years before screening (except for fully treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, localized prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery);
11. With severe liver function impairment:

    1. Total bilirubin ≥ 2.0 × upper limit of normal (ULN); for patients with Gilbert's syndrome, direct bilirubin ≥ 2.0 × ULN;
    2. Aspartate transaminase (AST) ≥ 5.0 × ULN, alanine transaminase (ALT) ≥5.0 × ULN;
12. With renal function impairment:

    1. Serum creatinine ≥2.0 × ULN;
    2. Creatinine clearance < 60 ml/min (calculated according to the Cockcroft-Gault formula, see Appendix 3 for details);
13. Pancreatic abnormalities:

    1. Serum amylase ≥ 2.0 × ULN;
    2. Serum lipase ≥ 2.0 × ULN;
14. More than 4 SBS or PN-related hospitalizations (such as catheter sepsis, intestinal obstruction, severe water and electrolyte disorders) within 12 months before screening;
15. Unplanned hospitalization within 30 days before screening;
16. Pregnant or lactating women, women or men who have fertility plans or do not agree to take effective contraceptive measures during the trial;
17. Participated in any clinical trial (excluding antibody treatment-related clinical trials) within 30 days before screening or participated in any antibody treatment-related clinical trials within 3 months before screening;
18. Other condition the investigator believes would be unsuitable for participation in this clinical study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of responders | Week 20 to 24 of treatment period
  A responder's PN/IV volume per week shows a reduction of at least 20% from baseline from week 20 to 24 in treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Huanlong Qin, Principal Investigator — Shanghai 10th People's Hospital
Locations (8):
- China (8):
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Xiangya Hospital of Central South University, Changsha, Hu'nan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No